CLINICAL TRIAL: NCT05787678
Title: Dupilumab Efficacy on Bronchial Inflammation, Small Airways Disfunction and Mucous Secretion in the Real Life Severe Asthma Patients
Brief Title: Dupilumab Efficacy on Bronchial Inflammation, Small Airways Disfunction and Mucous Secretion
Acronym: DEBORA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-DUP-2022-58
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-01

CONDITIONS: Asthma; Eosinophilic
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — dupilumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Induced sputum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Dupilumab — 600 mg (two 300 mg injections), followed by 300 mg monthly

SUMMARY:
Unicentric prospective real life study designed to analyse the efficacy of Dupilumab to reduce bronchial inflammation of asthma measured by inflammatory cell counts obtained in induced sputum and other related characteristics (small airway dysfunction and mucin production) in uncontrolled severe asthma patients in the real life setting without control group

DETAILED DESCRIPTION:
After patients signed informed consent, before (visit 1), after 4-5 months (visit 2), and after 12 months (visit 3) Dupilumab treatment began, the following techniques and measurements will be performed or collected: demographic data, blood analyses (eosinophil counts and total IgE), skin prick-test to common aeroallergens (only in the visit 1), asthma control test (ACT), sino-nasal outcome test (SNOT-22), test of adherence to inhalers (TAI), number of severe asthma exacerbations (in the previous year; in the visit 2, in the previous 4 months), oral and inhaled steroid daily doses received, spirometry, exhaled nitric oxide (FeNO), pulmonary volumes, carbon monoxide transference, oscillometry, and induced sputum (inflammatory cell counts and mucin profile [MUC1, MUC2, MUC5AC, MUC5B]). All patients will be performed at visits 1 and 3 in a 3D culture of primary nasal epithelial cells from asthmatic patients the pattern of gene and to identify new soluble biomarkers through quantitative proteomic analysis of culture supernatants.

Also a chest CT scan with expiratory images will be done only in visits 1 and 3.

ELIGIBILITY:
Inclusion Criteria:

* 18 -80 years
* Severe uncontrolled eosinophilic asthma by GINA (Global Initiative for Asthma) criteria
* Clinical indication of Dupilumab

Exclusion Criteria:

* Smoking over 10 pack/year
* Treatment with monoclonal antibodies treatment during the previous three months
* Refuse to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe uncontrolled eosinophilic asthma by GINA criteria with clinical indication of dupilumab
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of bronchial inflammatory cells | 1 year
  Count of induced sputum leucocytes

SECONDARY OUTCOMES:
Mucin production from epithelial cells | 1 year
  Levels of MUC 1, MUC2, MUC5AC, and MUC5B

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wenzel S, Castro M, Corren J, Maspero J, Wang L, Zhang B, Pirozzi G, Sutherland ER, Evans RR, Joish VN, Eckert L, Graham NM, Stahl N, Yancopoulos GD, Louis-Tisserand M, Teper A. Dupilumab efficacy and safety in adults with uncontrolled persistent asthma despite use of medium-to-high-dose inhaled corticosteroids plus a long-acting beta2 agonist: a randomised double-blind placebo-controlled pivotal phase 2b dose-ranging trial. Lancet. 2016 Jul 2;388(10039):31-44. doi: 10.1016/S0140-6736(16)30307-5. Epub 2016 Apr 27. PMID 27130691
- [Background] Castro M, Corren J, Pavord ID, Maspero J, Wenzel S, Rabe KF, Busse WW, Ford L, Sher L, FitzGerald JM, Katelaris C, Tohda Y, Zhang B, Staudinger H, Pirozzi G, Amin N, Ruddy M, Akinlade B, Khan A, Chao J, Martincova R, Graham NMH, Hamilton JD, Swanson BN, Stahl N, Yancopoulos GD, Teper A. Dupilumab Efficacy and Safety in Moderate-to-Severe Uncontrolled Asthma. N Engl J Med. 2018 Jun 28;378(26):2486-2496. doi: 10.1056/NEJMoa1804092. Epub 2018 May 21. PMID 29782217
- [Background] Rabe KF, Nair P, Brusselle G, Maspero JF, Castro M, Sher L, Zhu H, Hamilton JD, Swanson BN, Khan A, Chao J, Staudinger H, Pirozzi G, Antoni C, Amin N, Ruddy M, Akinlade B, Graham NMH, Stahl N, Yancopoulos GD, Teper A. Efficacy and Safety of Dupilumab in Glucocorticoid-Dependent Severe Asthma. N Engl J Med. 2018 Jun 28;378(26):2475-2485. doi: 10.1056/NEJMoa1804093. Epub 2018 May 21. PMID 29782224
- [Background] Wechsler ME, Ford LB, Maspero JF, Pavord ID, Papi A, Bourdin A, Watz H, Castro M, Nenasheva NM, Tohda Y, Langton D, Cardona G, Domingo C, Park HS, Chapman KR, Mao X, Zhang Y, Khan AH, Deniz Y, Rowe PJ, Kapoor U, Khokhar FA, Mannent LP, Ruddy M, Laws E, Amin N, Hardin M. Long-term safety and efficacy of dupilumab in patients with moderate-to-severe asthma (TRAVERSE): an open-label extension study. Lancet Respir Med. 2022 Jan;10(1):11-25. doi: 10.1016/S2213-2600(21)00322-2. Epub 2021 Sep 28. PMID 34597534
- [Background] Vega JM, Badia X, Badiola C, Lopez-Vina A, Olaguibel JM, Picado C, Sastre J, Dal-Re R; Covalair Investigator Group. Validation of the Spanish version of the Asthma Control Test (ACT). J Asthma. 2007 Dec;44(10):867-72. doi: 10.1080/02770900701752615. PMID 18097865
- [Background] Sanjuas C, Alonso J, Sanchis J, Casan P, Broquetas JM, Ferrie PJ, Juniper EF, Anto JM. [The quality-of-life questionnaire with asthma patients: the Spanish version of the Asthma Quality of Life Questionnaire]. Arch Bronconeumol. 1995 May;31(5):219-26. doi: 10.1016/s0300-2896(15)30927-3. Spanish. PMID 7788083
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] Plaza V, Alobid I, Alvarez C, Blanco M, Ferreira J, Garcia G, Gomez-Outes A, Gomez F, Hidalgo A, Korta J, Molina J, Pellegrini FJ, Perez M, Plaza J, Praena M, Quirce S, Sanz J. Spanish Asthma Management Guidelines (GEMA) VERSION 5.1. Highlights and Controversies. Arch Bronconeumol. 2022 Feb;58(2):150-158. doi: 10.1016/j.arbres.2021.05.010. Epub 2021 May 26. English, Spanish. PMID 34167859
- [Background] Garcia-Rio F, Calle M, Burgos F, Casan P, Del Campo F, Galdiz JB, Giner J, Gonzalez-Mangado N, Ortega F, Puente Maestu L; Spanish Society of Pulmonology and Thoracic Surgery (SEPAR). Spirometry. Spanish Society of Pulmonology and Thoracic Surgery (SEPAR). Arch Bronconeumol. 2013 Sep;49(9):388-401. doi: 10.1016/j.arbres.2013.04.001. Epub 2013 May 28. English, Spanish. PMID 23726118
- [Background] Paggiaro PL, Chanez P, Holz O, Ind PW, Djukanovic R, Maestrelli P, Sterk PJ. Sputum induction. Eur Respir J Suppl. 2002 Sep;37:3s-8s. doi: 10.1183/09031936.02.00000302. No abstract available. PMID 12361361
- [Background] Vidal S, Bellido-Casado J, Granel C, Crespo A, Plaza V, Juarez C. Flow cytometry analysis of leukocytes in induced sputum from asthmatic patients. Immunobiology. 2012 Jul;217(7):692-7. doi: 10.1016/j.imbio.2011.11.008. Epub 2011 Dec 2. PMID 22204819
- [Background] Pizzichini E, Pizzichini MM, Efthimiadis A, Evans S, Morris MM, Squillace D, Gleich GJ, Dolovich J, Hargreave FE. Indices of airway inflammation in induced sputum: reproducibility and validity of cell and fluid-phase measurements. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):308-17. doi: 10.1164/ajrccm.154.2.8756799.
- [Background] Magnussen H, Holz O, Sterk PJ, Hargreave FE. Noninvasive methods to measure airway inflammation: future considerations. Eur Respir J. 2000 Dec;16(6):1175-9. doi: 10.1034/j.1399-3003.2000.16f25.x. PMID 11292124
- [Background] Pepys J. Skin tests. Br J Hosp Med. 1984 Sep;32(3):120, 122, 124. PMID 6478105
- [Background] British Thoracic Society; Scottish Intercollegiate Guidelines Network. British guideline on the management of asthma. Thorax. 2014 Nov;69 Suppl 1:1-192. Epub 2014 Oct 16. No abstract available. PMID 25323740